CLINICAL TRIAL: NCT04659330
Title: Lipohypertrophy Monitoring Study
Acronym: LiMo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Principal Investigator, Christophe De Block, Professor, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17/41/458
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus; Lipohypertrophy; Hypoglycemia
Keywords: lipohypertrophy; online education; insulin injection technique; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Other): All patients underwent intervention
  Interventions: Behavioral: Online education (BdandMe) for injection technique; Device: 4mm needles

INTERVENTIONS:
Behavioral: Online education (BdandMe) for injection technique — patients were referred to the relevant modules on BD and Me™ (for online education)
Device: 4mm needles — Providing a supply of needles for single use of 4mm insulin injection needle.

SUMMARY:
The investigators intend to audit the impact of optimal injection technique education delivered through a multimodal tailored approach augmented with a digital 'tailorable' patient learning platform on clinical parameters and self-care behaviours of insulin treated patients in a prospective audit with follow-up in 6 months, conducted in multiple sites across Belgium. Diabetes patients with or without lipohypertrophy will be entered into the audit. The end points measured will include the impact on consumption of insulin, long term blood glucose control (HbA1c), hypoglycaemia, glucose variability, needle reuse, patient injection habits and clinician education, training and information inputs.

DETAILED DESCRIPTION:
Principle objective To assess the impact of optimal injection technique education, tailored learning prescription and use of BD Micro-FineTM Ultra 4mm x 32G pen needle upon total daily dose of insulin consumption in patients with or without clinically detectable lipohypertrophy. To assess the cost of intervention vs. direct savings with a view to use of the data in needle reimbursement discussions with the Belgian health care authorities.

Secondary objective

To assess the impact of the intervention on other parameters of glucose control (including HbA1c, unexplained hypoglycaemia and glycaemic variability). To calculate direct and indirect savings associated with better glucose control.

Tertiary objective

To assess the impact of the intervention (especially eLearning) on patients' injection technique self-care knowledge and behaviors, including correct site rotation, non-injection into lipohypertrophy and needle reuse patterns. To calculate direct and indirect savings associated with better educational approaches and behavioral changes.

Audit Targets and Standards The sample size targeted will be 190 completed patient records. Each center will be asked to contribute between 20-50 subjects. Optimal injection technique and optimal needle length selection are based on Belgian guidelines on Injection, which are based on recently published FITTER worldwide recommendations. A study day will be held for participant nurses to review the protocol and audit forms, and for refresher training in lipohypertrophy detection.

Endpoints Total Daily Dose (TDD) of insulin HbA1c (as mmol/mol) Unexplained hypoglycaemic episodes (defined in Entry/Exit Forms) Severe hypoglycaemia (requiring the intervention of a third party) Glycaemic variability (defined in Entry/Exit Forms) Rotation of injection sites with spacing apart of punctures by at least 1 cm Reuse of needles

Presence of lipohypertrophy Injections into lipohypertrophic lesions Injection technique practices Adherence to proposed best practice intervention recommendations Data with cost implications (resource usage, hypoglycaemic events) Self-care injection technique knowledge and behaviours Qualitative and quantitative BD and MeTM patient user experience Clinician education, training and information inputs required support behaviour modification and adherence to treatment Quality of Life assessment Unplanned Interventions: ER, Ambulance, Hospital Admission, Critical Cared admission

ELIGIBILITY:
Patient Inclusion Criteria

* Type 1 Diabetes Mellitus
* Type 2 Diabetes Mellitus
* Age 18 or above
* Injecting insulin for at least 1 year
* Self-managing injection therapy, including daily glucose monitoring
* Access to a device with internet
* Confident in navigating the internet

Patient Exclusion Criteria

* Children <18 years
* Pregnant or likely to become pregnant during study period
* Impaired cognitive ability which would prevent informed consent
* Syringe only user
* Insulin pump user
* GLP-1 RA therapy only
* Patients declining to take part in the study
* Cannot read and understand Dutch
* No access to an internet enabled device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Primary outcome parameter was the evolution between baseline and end-of-study percentage of needle reuse and injecting in a zone of lipohypertrophy.
Severe and unexplained hypoglycemia | 6 months
  Primary outcome parameter was the evolution between baseline and end-of-study percentage of needle reuse and injecting in a zone of lipohypertrophy.
  Hypoglycemia is defined as the occurrence of ≥ 1 symptom and a confirmed glucose reading ≤60 mg/dl. Unexplained hypoglycemia is defined as hypoglycemia occurring in the absence of a definable precipitating event such as a change in medication, diet or activity.
glucose variability | 6 months
  Primary outcome parameter was the evolution between baseline and end-of-study percentage of needle reuse and injecting in a zone of lipohypertrophy.
  Increased glucose variability was defined as the occurrence of at least 3 times a week glucose values evolving from <60 mg/dl (3.3 mmol/l) to >250 mg/dl (13.9 mmol/l) or vice versa (i.e. a delta >190 mg/dl or 10.6 mmol/l).

SECONDARY OUTCOMES:
Insulin dose in patients with and without lipohypertrophy | 6 months
  Secondary objectives were to evaluate the impact of the use of 4mm pen needles and an educational platform focused on correct injection technique, correct rotation of injection sites, non-injection into lipohypertrophy sites and stopping needle reuse on the insulin dose in patients with and without lipohypertrophy.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frid AH, Kreugel G, Grassi G, Halimi S, Hicks D, Hirsch LJ, Smith MJ, Wellhoener R, Bode BW, Hirsch IB, Kalra S, Ji L, Strauss KW. New Insulin Delivery Recommendations. Mayo Clin Proc. 2016 Sep;91(9):1231-55. doi: 10.1016/j.mayocp.2016.06.010. PMID 27594187
- [Background] Grassi G, Scuntero P, Trepiccioni R, Marubbi F, Strauss K. Optimizing insulin injection technique and its effect on blood glucose control. J Clin Transl Endocrinol. 2014 Jul 23;1(4):145-150. doi: 10.1016/j.jcte.2014.07.006. eCollection 2014 Dec. PMID 29159095
- [Background] Frid AH, Hirsch LJ, Menchior AR, Morel DR, Strauss KW. Worldwide Injection Technique Questionnaire Study: Injecting Complications and the Role of the Professional. Mayo Clin Proc. 2016 Sep;91(9):1224-30. doi: 10.1016/j.mayocp.2016.06.012. PMID 27594186
- [Background] Blanco M, Hernandez MT, Strauss KW, Amaya M. Prevalence and risk factors of lipohypertrophy in insulin-injecting patients with diabetes. Diabetes Metab. 2013 Oct;39(5):445-53. doi: 10.1016/j.diabet.2013.05.006. Epub 2013 Jul 22. PMID 23886784
- [Background] Ji L, Sun Z, Li Q, Qin G, Wei Z, Liu J, Chandran AB, Hirsch LJ. Lipohypertrophy in China: Prevalence, Risk Factors, Insulin Consumption, and Clinical Impact. Diabetes Technol Ther. 2017 Jan;19(1):61-67. doi: 10.1089/dia.2016.0334. PMID 28099050
- [Derived] Bochanen N, Decochez K, Heleu E, Cuypers J, Vercammen C, Coremans P, Vanhaverbeke G, Shadid S, Keymeulen B, Bolsens N, De Block C. Lipohypertrophy Monitoring Study (LIMO): Effect of single use of 4 mm pen needles combined with education on injection site rotation on glycaemic control: Confirmation of an unpleasant truth. Diabet Med. 2022 Jan;39(1):e14672. doi: 10.1111/dme.14672. Epub 2021 Sep 29. PMID 34407260